CLINICAL TRIAL: NCT06300645
Title: Split Tibialis Anterior Tendon Transfer to Peroneus Brevis vs Total Tibialis Anterior Tendon Transfer to Lateral Cuneiform in Recurrent Congenital Talipes Equinovarus: A Randomized Controlled Trial
Brief Title: SPLATT to Peroneus Brevis vs TATT to Lateral Cuneiform
Acronym: Recurrent CTEV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Yahya Abdelazeem Hassanein, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLATTvsTATT in recurrent CTEV
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Congenital Talipes Equinovarus
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPLATT (Experimental): Children with congenital talipes who have been treated with split tibialis anterior tendon transfer to peroneus brevis
  Interventions: Procedure: SPLATT
- TATT (Experimental): Children with congenital talipes who have been treated with total ribialis anterior tendon transfer to lateral cuneiform
  Interventions: Procedure: SPLATT

INTERVENTIONS:
Procedure: SPLATT — split tibialis anterior tendon transfer to peroneus brevis total tibialis anterior tendon transfer to lateral cuneiform
  Other Names: TATT

SUMMARY:
Congenital talipes equinovarus, is a common congenital foot deformity involving hindfoot equinus and varus, along with mid-/forefoot adduction and cavus. Currently, the Ponseti method is the preferred initial treatment for idiopathic clubfoot1

. Despite the initial phase's remarkable efficacy in correcting clubfeet, there remains a notable recurrence rate after Ponseti treatment2

* Numerous studies demonstrate a very high success rate during early follow-ups, ranging from 92% to 100%3
* Nonetheless, recurrence remains a challenge for orthopedic surgeons. A common trigger for recurrence is the dynamic supination of the foot, which results from excessive activation of the tibialis anterior muscle during ankle dorsiflexion4

Multiple studies indicate that tibialis anterior tendon transfer (TATT) is an effective tool for management of clubfoot recurrence, particularly dynamic supination5

* The widely used technique involves transferring the entire tendon through a drill hole in the lateral cuneiform and anchoring it on the plantar aspect of the foot using a sewing button and felt pad6
* While effective, this procedure raises the risk of pressure sores due to button placement on the sole7

Split anterior tibialis tendon transfer (SPLATT) to peroneus brevis is a well-described treatment strategy of varus foot deformities in patients with neuromuscular disorders8

* The technique has been reported to achieve successful deformity correction while avoiding skin problems associated with external button placement on the sole of the foot in tendon-to-bone transfers8

The present study aims to assess the outcome of utilizing SPLATT to peroneus brevis procedure in the treatment of recurrent CTEV in comparison to the original total TATT to the lateral cuneiform

ELIGIBILITY:
Inclusion Criteria:

* Recurrent CTEV
* Age between 4 years and 12 years
* Unilateral/bilateral
* Ankle dorsiflexion of at least 10° prior to tendon transfer

Exclusion Criteria:

* Non idiopathic CTEV
* Rigid deformity not suitable for acute correction
* Poor skin condition

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Correction of recurrent congenital talipes | 1 year
  correction is measured by arc of eversion

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt